CLINICAL TRIAL: NCT03563430
Title: Comparison of Acute Effects on Lactic Acid Removal, Flexibility, Strength, and Endurance of Different Recovery Methods
Brief Title: Effects of Different Recovery Methods on Lactic Acid Removal, Flexibility, Strength, and Endurance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Principal Investigator, Head of Physiotherapy and Rehabilitation Department, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BiruniU
Record Dates: First submitted 2018-05-28; First posted 2018-06-20 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Recovery Methods; Exercise Training
Keywords: foam roller; electrical stimulation; low intensity aerobic training; lactate removal

STUDY DESIGN:
Intervention Model Description: neuromuscular electrical stimulation, low intensity aerobic exercise, self massage with foam roller methods
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Recovery Group (Experimental): Participants in this group will exercise for 15 minutes, for a range of 65 to 70% of the maximum heart rate.
  Interventions: Other: Active Recovery Group
- Self-Massage with Foam Roller Group (Experimental): This group will perform 15 minutes self-massage with foam roller following the exercise session.
  Interventions: Other: Self-Massage with Foam Roller Group
- Neuromuscular Electrical Stimulation (Experimental): Participants of this group will be applied electrical stimulation on quadriceps femoris and hamstring muscles for 15 minutes while they are comfortable lying position.
  Interventions: Other: Neuromuscular Electrical Stimulation

INTERVENTIONS:
Other: Active Recovery Group — Participants in this group will exercise for 15 minutes, for a range of 65 to 70% of the maximum heart rate as a recovery method following a single bout high-intensity interval exercise program
  Arms: Active Recovery Group
Other: Self-Massage with Foam Roller Group — This group will perform 15 minutes self-massage with foam roller following the exercise session as a recovery method following a single bout high-intensity interval exercise program.
  Arms: Self-Massage with Foam Roller Group
Other: Neuromuscular Electrical Stimulation — Participants of this group will be applied electrical stimulation on quadriceps femoris and hamstring muscles for 15 minutes while they are comfortable lying position as a recovery method following a single bout high-intensity interval exercise program.
  Arms: Neuromuscular Electrical Stimulation

SUMMARY:
The aim of this study is to compare these three different recovery methods following a single bout high-intensity interval exercise program with each other in terms of blood lactate clearance, muscle flexibility, muscle strength and endurance.

DETAILED DESCRIPTION:
It is very important to choose the most effective recovery method for the athletes in training for their next training/competition. The recovery period is very significant in terms of removal of blood lactate and body dynamics as soon as they return to their original state and achieve high performance. Neither neuromuscular electrical stimulation, low-intensity aerobic exercise, self-massage with foam roller methods, which have been proven their effectiveness in the literature, have been compared with each other.

ELIGIBILITY:
Inclusion Criteria:

Young, healthy adults aged 20-25 years.

Exclusion Criteria:

* Clinical diagnosis of a cardiovascular disease.
* Clinical diagnosis of a metabolic disorder, orthopedic or neurological disease that would interfere with an exercise program,
* Clinical diagnosis of hemophili,
* Clinical diagnosis of thrombophlebitis or deep vein trombosis,
* Clinical diagnosis of peripheral arterial disease,
* Clinical diagnosis of venous insufficiency,
* Clinical diagnosis of anemia,
* Pregnancy.

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Blood Lactate change | change from baseline and 20. minutes of recovery
  blood lactate concentration measurement

SECONDARY OUTCOMES:
Quadriceps and Hamstring Muscle Strength | baseline and 1. hour
  Quadriceps and Hamstring Muscle Strength assessment with hand held dynamometer for left and right
Squat Endurance Test | baseline and 1. hour
  Squat endurance capacity assessment will done with 1 Repeat Maximum 60%
sit and reach test | baseline and 1. hour
  Hamstring Flexibility assessment will done with sit and reach test and will noted as centimeter

CONTACTS AND LOCATIONS:
Overall Officials: Buket AKINCI, PhD, Study Chair — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)